CLINICAL TRIAL: NCT01820104
Title: Effects of Lansoprazole on Sitagliptin Glucose-lowering Ability in Healthy Males
Brief Title: Effects of Lansoprazole on Sitagliptin Glucose-lowering Ability in Healthy Males: a Randomised Crossover Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20130301
Record Dates: First submitted 2013-03-17; First posted 2013-03-28 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — Lansoprazole; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): oral sitagliptin 100 mg on day 6 after administration of placebo (30 mg per day) for 6 days
- Combination of lansoprazole and sitagliptin (Experimental): oral sitagliptin 100 mg on day 6 after administration of lansoprazole (30 mg per day) for 6 days
  Interventions: Drug: lansoprazole, 30 mg per day for 6 days

INTERVENTIONS:
Drug: lansoprazole, 30 mg per day for 6 days
  Other Names: Oral glucose tolerance test (OGTT)
  Arms: Combination of lansoprazole and sitagliptin

SUMMARY:
Oral hypoglycemic medications sometimes do not control type 2 diabetes well. Proton pump inhibitors (PPIs) as adjunctive therapy might improve diabetes control and could enhance the hypoglycemic activity of DPP4, but there is little clinical data on efficacy of this therapeutic strategy. The investigators sought to examine the effect of PPI lansoprazole, DPP-4 inhibitor sitagliptin, and their combination therapy on insulin and glucose regulation in healthy subjects in oral glucose tolerance (OGTT).

DETAILED DESCRIPTION:
Oral hypoglycemic medications sometimes do not control type 2 diabetes well. Proton pump inhibitors (PPIs) as adjunctive therapy might improve diabetes control and could enhance the hypoglycemic activity of DPP4, but there is little clinical data on efficacy of this therapeutic strategy. We sought to examine the effect of PPI (lansoprazole), DPP4 (sitagliptin), and their combination therapy on insulin and glucose regulation in healthy subjects in oral glucose tolerance (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* General good health condition
* Male subject, between 18 and 50 years

Exclusion Criteria

* Overweight (Body Mass Index ≥30)
* Metabolic disorders
* History of gastrointestinal disorders
* Regular (daily) intake of medication
* Smoking more than 10 cigarettes/day
* History of drug abuse
* Exhaustive (> 3 units/day) alcohol consumption
* Exhaustive (> 5 units/day) caffeine consumption (coffee, tea, cola, or other caffeine based drinks)
* Recent (in the last 14 days) donation of blood
* Recent (in the last 2 days) donation of blood plasma
* Participation in another trial within 4 weeks before the start of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Glucose Tolerance | 0, 15, 30, 60, 90, 120, 180 min. after glucose administration

SECONDARY OUTCOMES:
Plasma insulin and C-peptide concentrations during oral glucose tolerance test | 0, 15, 30, 60, 90, 120, 180 min. after glucose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of pharmacy, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China